CLINICAL TRIAL: NCT05278429
Title: Robotic-assisted Exercise Training in Heart Failure With Reduced Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Heart Institute (Other)
Collaborators: ETH Zurich (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Myosuit Efficacy Trial
Record Dates: First submitted 2021-11-16; First posted 2022-03-14 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure, Systolic
Keywords: Exercise training; Robotic training
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myosuit arm (Active Comparator): Patients perform exercise training with the Myosuit
  Interventions: Device: Myosuit robotic device
- Control arm (Other): Patients perform exercise training without the Myosuit
  Interventions: Device: Myosuit robotic device

INTERVENTIONS:
Device: Myosuit robotic device — The Myosuit is a partially soft, exoskeleton-type, wearable robot that supports the synergistic extension of the hip and knee joints.

SUMMARY:
This study will address the challenging task of remobilizing patients with advanced chronic lung or heart failure in a functional New York Heart Association class III-IV by using an externally physically-supported exosuit movement therapy. This soft, wearable robot (Myosuit) assists mobilization according to individual needs by activating neuromuscular feedback systems, promoting physical activity and preventing early physical exhaustion.

The feasibility, tolerance and safety of a Myosuit assisted training was shown in a feasibility trial. In the efficacy trial, patients will be randomized in a 2:1 ratio for an exosuit-supported or non-supported exercise training protocol, training 3 units per week for 8 weeks. Assessment of outcome will be performed by various functional, mobility and endurance tests, questionnaires and clinical parameters. Furthermore, the transfer of regained motor and balance skills to everyday life will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* >17 years old
* written informed consent
* chronic end-stage systolic heart failure without ventricular assist device, LVEF ≤ 45%
* clinically stable for at least 6 weeks
* ability to mobilize into standing and walking of at least 10 meters with or without rollator
* ability to get up from a chair without rotating the upper body >45° sagittally

Exclusion Criteria:

* addictions or other illnesses that impact the ability to understand the nature, scope and
* consequences of the trial
* lack of knowledge of German to fully understand study information
* pregnancy, pre-menopausal women
* contraindications of cardiopulmonary exercising
* BMI > 35 kg/m², waist size > 135 cm.
* Height <150 cm, >195 cm
* Weight<45 kg, >110 kg
* Functional Reach Test <15,24 cm
* Flexion contracture in the knee/hip joint >10°
* Chronic colonization or active infection with multi-resistant pathogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity improves more in patients who trained with robotic support | 8 weeks
  Exercise capacity is measured by six-minute walking test in meters
Exercise capacity improves more in patients who trained with robotic support | 4 weeks
  Exercise capacity is measured by six-minute walking test in meters
Mobility improves more in patients who trained with robotic support | 8 weeks
  Mobility is measured by timed-up-and-go tests in seconds
Mobility improves more in patients who trained with robotic support | 4 weeks
  Mobility is measured by timed-up-and-go tests in seconds
Balance improves more in patients who trained with robotic support | 8 weeks
  Balance is measured by berg balance tests via berg balance scale (0-56 points, the higher, the better).
Balance improves more in patients who trained with robotic support | 4 weeks
  Balance is measured by berg balance tests via berg balance scale(0-56 points, the higher, the better).
Exercise training improves quality of life | 8 weeks
  Quality of life is measured by Kansas City Cardiomyopathy Questionnaire
Heart failure Progression: Ejection fractions | 4 weeks
  Change of echocardiographic findings: ejection fraction (in %)
Heart failure Progression: Diameters | 8 weeks
  Change of echocardiographic findings: diameters (in mm)
Heart failure Progression: valve regurgitations | 8 weeks
  Change of echocardiographic findings: regurgitations (grad I-V)
Heart failure Progression: elevated filling pressures | 8 weeks
  Change of echocardiographic findings: end-diastolic pressure (elevated or normal)
Heart failure Progression: volume status | 8 weeks
  Change of echocardiographic findings: vena cava diameter (in mm)
Change in Heart failure biomarkers: NT-proBNP | 8 weeks
  Heart failure biomarkers: NT-proBNP
Change in Heart failure biomarkers: hsTroponin | 8 weeks
  Heart failure biomarkers: hsTroponin
Change in inflammatory biomarkers: hsCRP | 8 weeks
  Inflammatory biomarkers: NT-proBNP (in ng/mL)
Change in inflammatory biomarkers: IL-6 | 8 weeks
  Inflammatory biomarkers: IL-6

SECONDARY OUTCOMES:
Device acceptability | 8 weeks
  measured by a acceptability questionnaire (9 questions, Score 9 to 63, the higher, the better).

CONTACTS AND LOCATIONS:
Locations (1):
- German Heart Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No